CLINICAL TRIAL: NCT03481010
Title: Periacetabular Osteotomy With and Without Arthroscopic Management of Central Compartment Pathology: A Multicenter Randomized Controlled Trial
Brief Title: Periacetabular Osteotomy With and Without Arthroscopic Management of Central Compartment Pathology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170796
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation | interventions — Polyamine Oxidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAO with hip arthroscopy (Experimental): Patient's in the "Scope PAO" group have been diagnosed with hip dysplasia and a decision has been made between the patient and the surgeon that the best way to treat the hip problems is with surgery. Patient's in the "Scope-PAO" group have been randomized to receive a periacetabular osteotomy with a hip arthroscopy.
  Interventions: Procedure: PAO with hip arthroscopy
- PAO without hip arthroscopy (Active Comparator): Patient's in the "PAO-only" group have been diagnosed with hip dysplasia and a decision has been made between the patient and the surgeon that the best way to treat the hip problems is with surgery. Patient's in the "PAO-only" group have been randomized to receive a periacetabular osteotomy only.
  Interventions: Procedure: PAO without hip arthroscopy

INTERVENTIONS:
Procedure: PAO with hip arthroscopy — Participants who are randomized to the Scope-PAO group will receive central compartment hip arthroscopy in addition to the PAO.
  Arms: PAO with hip arthroscopy
Procedure: PAO without hip arthroscopy — Participants who are randomized to the "PAO-only" group will receive a Bernese Periacetabular Osteotomy (PAO) for treatment of hip dysplasia.
  Arms: PAO without hip arthroscopy

SUMMARY:
At present, it is not clear whether performing a hip arthroscopy at the same time as a PAO improves patient outcomes after surgery compared to a PAO alone.

This research project will randomize patients to receive either a PAO alone, or a PAO and a hip arthroscopy at the same time.

DETAILED DESCRIPTION:
Hip dysplasia is a developmental abnormality of the acetabulum (hip socket) that causes abnormal stresses inside the hip joint and leads to painful arthritis at a young age. Many patients develop painful symptoms in their hip before advanced arthritis occurs.

The periacetabular osteotomy (PAO) is a surgical procedure that reorients the acetabulum to reduce the stresses inside the hip joint. The PAO is very effective at improving symptoms and quality of life. However, some patients may have residual symptoms.

Frequently, people with hip dysplasia will have an MRI done before their surgery, which helps to identify other the abnormalities inside their hip joint (e.g., labral tears). These abnormalities inside the joint cannot easily be addressed through PAO alone, however they can be addressed with hip arthroscopy. Hip arthroscopy is a separate minimally invasive surgical procedure that allows the surgeon to access the inside of the hip joint with a small camera and address any abnormalities.

At present, it is not clear whether performing a hip arthroscopy at the same time as a PAO improves patient outcomes after surgery compared to a PAO alone.

This research project will randomize patients to receive either a PAO alone, or a PAO and a hip arthroscopy at the same time. Patients will be followed for 2 years after surgery. Symptomatic differences between the two patient groups will be assessed to determine added benefit of the hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patient undergoing Bernese periacetabular osteotomy for symptomatic acetabular dysplasia/hip instability
* Pre-Operative MRI at 3T and/or gadolinium MR arthrogram
* Age, 16-50 years old
* Patient capable of giving informed consent

Exclusion Criteria:

* Prior hip/pelvis surgery of any kind on the surgical side
* Prior hip arthroplasty surgery on either side
* Radiographic evidence of arthritis (i.e. Tönnis grade =2)
* Known connective tissue disorder (e.g. Ehlers-Danlos Syndrome, etc.)
* Known neuromuscular disorder (e.g. Cerebral Palsy, Spina bifida, etc.)
* Known skeletal dysplasia (e.g. Achondroplasia, Multiple Epiphyseal Dysplasia, etc.)
* Cognitive impairment that prevents accurate completion of patient-reported outcome questionnaires.
* Patient unable/unwilling to complete all required follow-up visits
* Concurrent proximal femoral osteotomy and/or surgical hip dislocation

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
iHOT-33 | 24 months
  Patient-reported quality of life will be the primary outcome used for comparison between the two treatment groups as measured by the International Hip Outcome Tool (iHOT-33). The iHOT-33 is a validated, self-administered quality of life assessment tool for young, active patients with hip symptoms.

SECONDARY OUTCOMES:
HOOS | before surgery, 6 months, 12 months, 24 months after surgery
  Hip-specific symptoms and functional impairment will be compared using the Hip Disability and Osteoarthritis Outcome Score (HOOS). This 40-item patient reported outcome tool has been validated for use in patients with and without hip osteoarthritis and has shown good responsiveness, reliability and reproducibility in this patient population.
PROMIS Global 10 | before surgery, 6 months, 12 months, 24 months after surgery
  Global Health assessment will be compared using the PROMIS Global 10 Score. This 10-item tool assesses general domains of health related quality of life in the domains of physical, mental, and social well-being.
Operative time | intra-operative
  Total operative time is expected to be longer in the "Scope-PAO" treatment group, however the average increase in time will be valuable information for future research assessing cost-effectiveness of this treatment strategy. Total operative time will be measured from the time the patient enters the operating room to the time the patient is ready for transfer to post-anesthetic care unit (PACU). This time interval represents the best assessment of the overall time cost to the health care system associated with the surgical procedure while avoiding confounding due to delays in transfer to PACU.
Hospital Length of Stay | up to one month
  Length of stay, measured in days, will be assessed from date of admission to date of discharge up to one month.
Adverse Events | 2-4 weeks and 3 months after surgery
  Adverse events will be assessed prospectively at the first and second post-operative visits using Sink et al.'s classification system that grades the complications based on required treatment and long-term morbidity.
Cost-Effectiveness | 6 months, 12 months, and 24 months after surgery
  The cost-effectiveness of the two study groups will be assessed prospectively using the Work Productivity and Activity Impairment Questionnaire. This 6-item validated questionnaire quantifies work impairments. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism and percentage of impairment in activities performed outside of work. Greater scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Wilkin, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (7):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - The Washington University, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
- Canada (3):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - CHU de Québec - Université Laval, Québec

REFERENCES:
- [Derived] Wilkin GP, Poitras S, Clohisy J, Belzile E, Zaltz I, Grammatopoulos G, Melkus G, Rakhra K, Ramsay T, Thavorn K, Beaule PE. Periacetabular osteotomy with or without arthroscopic management in patients with hip dysplasia: study protocol for a multicenter randomized controlled trial. Trials. 2020 Aug 18;21(1):725. doi: 10.1186/s13063-020-04592-9. PMID 32811527